CLINICAL TRIAL: NCT01584557
Title: A Phase 3 Randomized, Double-Blind, Placebo Controlled Study of the Short Term Clinical Effects of Tolvaptan in Patients Hospitalized for Worsening Heart Failure With Challenging Volume Management
Brief Title: Randomized, Double-Blind, Placebo Controlled Study of the Short Term Clinical Effects of Tolvaptan in Patients Hospitalized for Worsening Heart Failure With Challenging Volume Management
Acronym: Secret of CHF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cardiovascular Clinical Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCSF-2011-001
Record Dates: First submitted 2012-04-10; First posted 2012-04-25 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan, Samsca (Active Comparator): Tolvaptan, Samsca, uncoated tablet, 30 mg, once per day, up to 7 days.
  Interventions: Drug: Tolvaptan or Samsca
- sugar pill (Placebo Comparator): placebo, sugar pill
  Interventions: Drug: placebo or sugar pill

INTERVENTIONS:
Drug: Tolvaptan or Samsca — uncoated tablet, 30mg, once per day, for up to 7 days.
  Arms: Tolvaptan, Samsca
Drug: placebo or sugar pill — sugar pill
  Arms: sugar pill

SUMMARY:
The purpose of this study is to evaluate the short term efficacy and safety of tolvaptan in subjects hospitalized for worsening heart failure who have volume overload and one of the following: renal insufficiency, or hyponatremia or inadequate response to diuretic therapy. The primary variable for assessing efficacy will be self-assessed 7-point dyspnea score at 8 and 16 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects hospitalized for worsening heart failure and randomized within 36 hours of initial presentation.
2. Males and females 18 years of age or older.
3. NYHA Class III or IV on admission to the hospital.
4. Able to understand content of and willing to provide written informed consent
5. Dyspnea, measured by the 5-point current dyspnea scale (moderately short of breath or worse), within 2 hours of randomization and dosing.

   The following must be met within 12 hours of randomization.
6. The subject must have signs of extracellular volume expansion, defined as two or more of the following five: Signs of RHF ( jugular venous distention, pitting edema (≥1+), ascites) and/or Signs of LHF (pulmonary congestion on chest x-ray, pulmonary rales)
7. Have at least one of the following:

   * eGFR < 60ml/min/1.73m2, OR
   * serum sodium ≤ 134 mEq/L, OR
   * urine output ≤ 125 ml/hr over anytime frame of at least 2 hours, following administration of IV furosemide of at least 40mg. See table below.

Time Period (hr) Cumulative UO (mL) 2 <250 3 <375 4 <500 5 <625 6 <750 7 <875 8 <1000

Exclusion Criteria:

1. Positive urine pregnancy test for women of child bearing potential.
2. Inability to provide written informed consent.
3. Cardiac surgery within 60 days prior to study randomization.
4. Acute Coronary Syndrome (ACS) or percutaneous coronary intervention within 30 days prior to study randomization.
5. Planned revascularization procedures, cardiac mechanical support implantation, cardiac transplantation, or other cardiac surgery within 30 days following study randomization.
6. Planned electrophysiologic (EP) device implantation within 7 days following study randomization.
7. Subjects who are on cardiac mechanical support.
8. Co-morbid condition with an expected survival less than six months.
9. History of a cerebrovascular accident within the last 30 days.
10. Hemodynamically significant uncorrected primary cardiac valvular disease.
11. Hypertrophic cardiomyopathy (obstructive or non-obstructive).
12. Uncorrected thyroid disease, active myocarditis or known amyloid cardiomyopathy.
13. History of primary significant liver disease or acute hepatic failure, as defined by the investigator.
14. Chronic uncontrolled diabetes mellitus as determined by the investigator.
15. Supine systolic arterial blood pressure < 90 mmHg.
16. Serum creatinine > 3.5 mg/dL or undergoing dialysis.
17. Hemoglobin < 9 g/dL
18. History of hypersensitivity and/or idiosyncratic reaction to benzazepine derivatives (such as benazepril).
19. Inability to take oral medications.
20. Participation in another clinical drug or device trial where the last dose of drug was within the past 30 days or an investigational medical device is currently implanted.
21. Previous exposure to tolvaptan within 7 days prior to randomization.
22. Subjects with refractory, end-stage, heart failure defined as subjects who are appropriate candidates for specialized treatment strategies, such as ventricular assist devices, continuous positive IV inotropic therapy, or hospice care.
23. Ultrafiltration within 7 days prior to randomization or planned.
24. Active gout
25. Serum sodium >144 mEq/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the short term efficacy and safety of tolvaptan in subjects hospitalized for worsening heart failure who have volume overload and one of the following: renal insufficiency, or hyponatremia or inadequate response to diuretic therapy. | 8 and 16 hours
  The primary variable for assessing efficacy will be self-assessed 7-point dyspnea score at 8 and 16 hours.

SECONDARY OUTCOMES:
Change from baseline in body weight measured daily while hospitalized up to 7 days. | up to 7 days
  Change from baseline in body weight measured daily while hospitalized up to 7 days.
Diuretic dose measured daily while hospitalized up to 7 days. | up to 7 days.
  Diuretic dose measured daily while hospitalized up to 7 days.
Change from baseline in estimated glomerular filtration rate (eGFR) at discharge or day 7, whichever comes first. | at discharge or day 7, whichever comes first.
  Change from baseline in estimated glomerular filtration rate (eGFR) at discharge or day 7, whichever comes first.
Days alive and out of the hospital over 30 days | 30 days.
  Days alive and out of the hospital over 30 days
Change from baseline in cognitive function at 48 hours or discharge, whichever comes first | at 48 hours or dischage, whichever comes first
  Change from baseline in cognitive function at 48 hours or discharge, whichever comes first
Re-hospitalization for worsening heart failure or death at 30 days | 30 days.
  Re-hospitalization for worsening heart failure or death at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Konstam, MD, Principal Investigator — Cardiovascular Clinical Sciences Inc
Locations (37):
- United States (37):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Heart Center Research, Huntsville, Alabama
  - Greater Los Angeles VA Medical Center, Los Angeles, California
  - University of Florida Health Science Ctr. Jacksonville, Jacksonville, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University Cardiology Associates, LLC, Augusta, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Advocate Medical Group - Oakbrook, Naperville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - CardioSpecialists Group, Munster, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - Louisiana Heart Center and Research, Slidell, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Crittenton Hospital Medical Center, Rochester, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Bryan Heart Institute, Lincoln, Nebraska
  - The Valley Hospital, Ridgewood, New Jersey
  - Caromont Heart/Gaston Memorial Hospital, Gastonia, North Carolina
  - Duke Cardiology of Lumberton Research/Southeastern Regional Medical Cente, Lumberton, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - University of Cincinnati, Cincinnatti, Ohio
  - Dayton Heart Center, Dayton, Ohio
  - The Sisters of Mercy of Hamilton, Ohio dba Mercy Hospital Fairfield, Fairfield, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Memorial Hospital of RI, Pawtucket, Rhode Island
  - The Miriam Hosptial, Providence, Rhode Island
  - University of Texas Health Science Center, Houston, Texas
  - The Heart Hospital Baylor Plano - Research Insititute, Plano, Texas
  - CV Group Central Lynchburg/Stroobants Heart Center, Lynchburg, Virginia
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Konstam MA, Kiernan M, Chandler A, Dhingra R, Mody FV, Eisen H, Haught WH, Wagoner L, Gupta D, Patten R, Gordon P, Korr K, Fileccia R, Pressler SJ, Gregory D, Wedge P, Dowling D, Romeling M, Konstam JM, Massaro JM, Udelson JE; SECRET of CHF Investigators, Coordinators, and Committee Members. Short-Term Effects of Tolvaptan in Patients With Acute Heart Failure and Volume Overload. J Am Coll Cardiol. 2017 Mar 21;69(11):1409-1419. doi: 10.1016/j.jacc.2016.12.035. PMID 28302292